CLINICAL TRIAL: NCT05716204
Title: Effects on Pain, Strength and Functional Capacity of High Force Distraction of the Hip in Athletes With Osteitis Pubis.
Brief Title: Effects of Manual Therapy in Strenght, Pain and Functional Capacity for Sport Related Groin Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This record was created in error.
Sponsor: University of Valladolid (Other)
Responsible Party: Principal Investigator, Silvia Lahuerta Martín, Principal investigator, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 067/229211
Record Dates: First submitted 2023-01-16; First posted 2023-02-08 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2023-11

CONDITIONS: Osteitis Pubis; Athletic Pubalgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High force lateral distraction group (Experimental): High force lateral distraction of the hip in maximun adjusted position.
  Interventions: Other: High force lateral distraction
- Placebo distraction group (Sham Comparator): Placebo lateral distraction of the affected hip in maximun adjusted position.
  Interventions: Other: Placebo distraction group

INTERVENTIONS:
Other: High force lateral distraction — High force lateral distraction on the affected hip.
  Arms: High force lateral distraction group
Other: Placebo distraction group — Placebo lateral distraction on the affected hip.
  Arms: Placebo distraction group

SUMMARY:
Athletic osteitis pubis is a pathologic entity that can cause functional impairment. Scientific evidence have noticed that athletes experiment pain and a decrease on strength. Moreover, this symptomathology can affect daily life and functionality. There is no scientific evidence about the influence of manual therapy (MT) as a single treatment to improve this condition. The investigators decided to conduct a randomized controlled trial to compare the effects of a MT technique with placebo technique.

ELIGIBILITY:
Inclusion Criteria:

* Athletes diagnosed with osteitis pubis stage 1 with at least 3 months of evolution.
* Internal rotation ROM limited.
* Positive provocation pain tests.

Exclusion Criteria:

* Pain due to intraarticular hip pathology.
* Hip pain due to inflamatory diseases.
* Previous surgical interventions in hip, pelvis or lumbar spine.
* MRI results or provocation pain tests inconcluyent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Strength | Baseline
  Strength evaluate for internal and external hip rotators with a conical pulley.
Strength | Through study completion, an average of two weeks
  Strength evaluate for internal and external hip rotators with a conical pulley.
Strength | 3 months follow-up
  Strength evaluate for internal and external hip rotators with a conical pulley.

SECONDARY OUTCOMES:
Pain in sports activities | Baseline
  Appearance time of pain during activities
Pain in sports activities | Through study completion, an average of two weeks
  Appearance time of pain during activities
Pain in sports activities | 3 months follow-up
  Appearance time of pain during activities
Pain intensity during/after pain provocation tests: Single adductor, squeeze and bilateral adductor tests | Baseline
  Appearance of pain during or after the execution of Single adductor, squeeze and bilateral adductor tests. If pain appears it will be reported by the patient using visual analog scale (VAS) from 0 to 10, in which higher scores are worse.
Pain intensity after pain provocation tests: Single adductor, squeeze and bilateral adductor tests | Through study completion, an average of two weeks
  Appearance of pain during or after the execution of Single adductor, squeeze and bilateral adductor tests. If pain appears it will be reported by the patient using visual analog scale (VAS) from 0 to 10, in which higher scores are worse.
Pain intensity after pain provocation tests: Single adductor, squeeze and bilateral adductor tests | 3 months follow-up
  Appearance of pain during or after the execution of Single adductor, squeeze and bilateral adductor tests. If pain appears it will be reported by the patient using visual analog scale (VAS) from 0 to 10, in which higher scores are worse.
Functional capacity | Baseline
  Evaluated with a patient reported outcome questionnaire called Copenhagen Hip and Groin Outcome score (HAGOS) which assesses pain, symptoms, physical function in daily living, physical function in sport and recreation, participation in physical activities and hip and groin -related quality of life. For each item answer range from "never" to "always".
Functional capacity | Through study completion, an average of two weeks
  Evaluated with a patient reported outcome questionnaire called Copenhagen Hip and Groin Outcome score (HAGOS) which assesses pain, symptoms, physical function in daily living, physical function in sport and recreation, participation in physical activities and hip and groin -related quality of life. For each item answer range from "never" to "always".
Functional capacity | 3 months follow-up
  Evaluated with a patient reported outcome questionnaire called Copenhagen Hip and Groin Outcome score (HAGOS) which assesses pain, symptoms, physical function in daily living, physical function in sport and recreation, participation in physical activities and hip and groin -related quality of life. For each item answer range from "never" to "always".

OTHER OUTCOMES:
Treatment expectancy and credibility | Through study completion, an average of two weeks
  Evaluated with Credibility and expectancy Questionaire (CEQ) in which the patient answer question related to the expectations of the intervention. Higher values mean better expectations on the therapy.
Treatment expectancy and credibility | 3 months follow-up
  Evaluated with Credibility and expectancy Questionaire (CEQ) in which the patient answer question related to the expectations of the intervention. Higher values mean better expectations on the therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Lahuerta Martín, Principal Investigator — University of Valladolid; Luis Ceballos Laita, Study Director — University of Valladolid; Sandra Jiménez del Barrio, Study Director — University of Valladolid; Maria Teresa Mingo Gómez, Study Director — University of Valladolid
Locations (1):
- Silvia Lahuerta Martín, Soria, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verrall GM, Slavotinek JP, Barnes PG, Fon GT. Description of pain provocation tests used for the diagnosis of sports-related chronic groin pain: relationship of tests to defined clinical (pain and tenderness) and MRI (pubic bone marrow oedema) criteria. Scand J Med Sci Sports. 2005 Feb;15(1):36-42. doi: 10.1111/j.1600-0838.2004.00380.x. PMID 15679570
- [Background] Thorborg K, Holmich P, Christensen R, Petersen J, Roos EM. The Copenhagen Hip and Groin Outcome Score (HAGOS): development and validation according to the COSMIN checklist. Br J Sports Med. 2011 May;45(6):478-91. doi: 10.1136/bjsm.2010.080937. PMID 21478502
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119